CLINICAL TRIAL: NCT03587090
Title: Comparaison échographique Des Voies Sous Costale et Trans hépatique Dans l'évaluation de la Veine Cave inférieure
Brief Title: Comparison of Subcostal and Transhepatic Views to Assess Inferior Vena Cava by Echocardiography
Acronym: VCI ECHO
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: caenUH 18-034
Record Dates: First submitted 2018-06-08; First posted 2018-07-16 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-06

CONDITIONS: Inferior Vena Cava Diameter
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echocardiography — echocardiography by subcostal and transhepatic views

SUMMARY:
Comparison of subcostal and transhepatic views to measure inferior vena cava diameter by echocardiography in intensive care unit patients

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalised in ICU

Exclusion Criteria:

* gardianship
* contraindication to transthoracic echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
inferior vena cava diameter | up to 1 day after inclusion
  measurement of inferior vena cava diameter by 2D et TM mode

CONTACTS AND LOCATIONS:
Locations (1):
- Service de réanimation médicale CHU de Caen, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided